CLINICAL TRIAL: NCT02967510
Title: A Phase 2, Dose-ranging, 12-week Randomized, Double-blind, Placebo Controlled, Parallel-group Study Evaluating the Efficacy and Safety of Three Formulations of Ultra-low Dose Estriol Vaginal Gel (0.005% Estriol Vaginal Gel, 0.002% Estriol Vaginal Gel, 0.0008% Estriol Vaginal Gel) for the Treatment of Vaginal Dryness in Postmenopausal Women With Vulvovaginal Atrophy
Brief Title: Study Evaluating the Efficacy and Safety of Three Formulations of Ultra-low Dose Estriol Vaginal Gel (0.005%, 0.002%, 0.0008% Estriol Vaginal Gel) for the Treatment of Vaginal Dryness in Postmenopausal Women With Vulvovaginal Atrophy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: ITF Research Pharma, S.L.U. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ITFE-2092-C1; 2015-005787-42 (EudraCT Number)
Record Dates: First submitted 2016-11-11; First posted 2016-11-18 (Estimated); Results first posted 2019-09-25 (Actual); Last update posted 2019-09-25 (Actual); Status verified 2019-08

CONDITIONS: Vaginal Atrophy
MeSH Terms: interventions — Estriol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- 0.005% estriol vaginal gel (Experimental): Vaginal. Administration by an applicator inserted deep inside the vagina Dose: 1 g of gel, containing 50 Mcg of estriol Dosage schedule: Weeks 1-3: single daily application Weeks 4-12: twice weekly administration
  Interventions: Drug: Estriol
- 0.002% estriol vaginal gel (Experimental): Vaginal. Administration by an applicator inserted deep inside the vagina Dose: 1 g of gel, containing 50 Mcg of estriol Dosage schedule: Weeks 1-3: single daily application Weeks 4-12: twice weekly administration
  Interventions: Drug: Estriol
- 0.0008% estriol vaginal gel (Experimental): Vaginal. Administration by an applicator inserted deep inside the vagina Dose: 1 g of gel, containing 50 Mcg of estriol Dosage schedule: Weeks 1-3: single daily application Weeks 4-12: twice weekly administration
  Interventions: Drug: Estriol
- estriol vaginal gel (Placebo Comparator): Vaginal. Administration by an applicator inserted deep inside the vagina Dose: 1 g of gel, containing 50 Mcg of estriol Dosage schedule: Weeks 1-3: single daily application Weeks 4-12: twice weekly administration
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Estriol
  Arms: 0.0008% estriol vaginal gel; 0.002% estriol vaginal gel; 0.005% estriol vaginal gel
Drug: Placebo
  Arms: estriol vaginal gel

SUMMARY:
A Phase 2, Dose-ranging, 12-week Randomized, Double-blind, Placebo controlled, Parallel-group Study Evaluating the Efficacy and Safety of Three Formulations of Ultra-low Dose Estriol Vaginal Gel (0.005% Estriol Vaginal Gel, 0.002% Estriol Vaginal Gel, 0.0008% Estriol Vaginal Gel) for the Treatment of Vaginal Dryness in Postmenopausal Women with Vulvovaginal Atrophy.

Vulvovaginal atrophy is a natural consequence of the progressive estrogen deficiency that occurs in menopause. Epidemiological data have indicated that about 50% of otherwise healthy women over 60 years of age experience symptoms related to urogenital atrophy such as vaginal dryness, dyspareunia, burning, itching, as well as urinary complaints or infections of the lower urinary tract. As these alterations frequently affect the quality of life of postmenopausal women, it is important for doctors to detect their presence and offer treatment options. Estrogen therapy is the most effective treatment of moderate to severe symptoms of vulvar and vaginal atrophy. One advantage of local treatment with estrogen is avoidance of first-pass liver metabolism, making it possible to use lower doses of estrogen compared with oral therapy; the local route also minimize systemic adverse effects. The search for therapeutic alternatives which may present improvements in relation to the current products has been encouraged.

ELIGIBILITY:
Inclusion Criteria:

1. Capable of understanding the written informed consent, provides signed and witnessed written informed consent, and agrees to comply with the protocol procedures and assessments
2. Age >40 and <80 years
3. Postmenopausal (≥12 months since last spontaneous menstrual period, or having 6 months of spontaneous amenorrhea with serum FSH levels >40 IU/L, or ≥6 weeks since bilateral oophorectomy with or without hysterectomy)
4. BMI ≤36 kg/m2
5. Vaginal Maturation Index ≤ 5% superficial cells on a vaginal smear
6. Vaginal pH >5
7. Moderate to severe vaginal dryness currently reported as the most bothersome symptom of vaginal atrophy.
8. Documented negative mammogram within 9 months prior to randomization, with normal breast examination at screening.
9. Negative Papanicolau test at screening (in women with cervix).

Exclusion Criteria:

1. Subjects with contraindications for hormone therapy with estrogens such as those diagnosed or history of: malignant and premalignant lesions of the breast and/or endometrium, malignancy of the colon, malignant melanoma, hepatic tumor, venous thromboembolic conditions (including deep vein thrombosis or pulmonary embolism), arterial thromboembolic conditions (including angina pectoris, myocardial infarction, or cerebrovascular accident), coagulopathies, vaginal bleeding of unknown etiology, acute liver disease or a history of liver disease as long as liver function tests have failed to return to normal, or porphyria.
2. Subjects who have abnormal laboratory values at screening that the investigator considers clinically relevant for the purposes of the study.
3. Subjects with any medical-surgical pathology which is not controlled at the time of inclusion in the study
4. Subjects with any acute or chronic condition whose management or progression may interfere with the subject´s participation in the study.
5. Subject with uncontrolled hypertension (>140 mmHg systolic blood pressure and/or ≥90 mmHg diastolic blood pressure).
6. Subjects with Grade II or higher utero-vaginal prolapse.
7. Subjects with uterine polyps.
8. Subjects with symptomatic and/or large uterine fibroids (>3 cm) and/or palpable fibroids at gynecological examination.
9. Subjects who have had urogenital surgery within 3 months of baseline visit.
10. Subjects with signs and symptoms suggestive of infection of the genital or urinary tract requiring treatment at the start of the study.
11. In women who have a uterus, evidence of hyperplasia, cancer or other endometrial pathology in endometrial biopsy.
12. Subjects who have received the following treatments within the specified time periods prior to screening procedures: any type of non-hormonal vulvovaginal treatment in the 7 days (including cosmetics expected to have an impact on vaginal pH such as special feminine wash gels); phytoestrogens by any route within 1 month; vaginal hormone therapy within 1 month; hormone therapy (estrogen alone, progestin alone or estrogen/progestin combination) by oral, intrauterine or transdermal route within 2 months; progestational implants, estrogen, or estrogen/progestational injectable within 3 months; estrogen pellet therapy or progestin injectable drug therapy within 6 months; percutaneous estrogen lotions or gels within 1 month; testosterone or testosterone derivatives, DHEA, tibolone, or SERMs by any route within 2 months;
13. Subjects receiving antiepileptic drugs (barbiturates, hydantoins, carbamazepine), certain antibiotics and other antiinfective medicinal products; phenylbutazone; preparations based on medicinal plants that contain St. John's Wort.
14. Subjects who are allergic to any of the components of the medication under study.
15. Subjects who are currently participating or have participated in the experimental evaluation of any product within 8 weeks of the start of the study

Ages: 40 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 283 (Actual)
Dates: Start 2016-10; Primary Completion 2018-05 (Actual); Study Completion 2018-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (22):
- Czechia (6):
  - For additional information regarding investigative sites for this trial, contact ITF Research Pharma S.L.U, Brno
  - For additional information regarding investigative sites for this trial, contact ITF Research Pharma S.L.U., České Budějovice
  - For additional information regarding investigative sites for this trial, contact ITF Research Pharma S.L.U., Olomouc
  - For additional information regarding investigative sites for this trial, contact ITF Research Pharma S.L.U., Písek
  - For additional information regarding investigative sites for this trial, contact ITF Research Pharma S.L.U., Prague
  - For additional information regarding investigative sites for this trial, contact ITF Research Pharma S.L.U., Vsetín
- Hungary (4):
  - For additional information regarding investigative sites for this trial, contact ITF Research Pharma S.L.U, Szeged
  - For additional information regarding investigative sites for this trial, contact ITF Research Pharma S.L.U., Szentes
  - For additional information regarding investigative sites for this trial, contact ITF Research Pharma S.L.U, Székesfehérvár
  - For additional information regarding investigative sites for this trial, contact ITF Research Pharma S.L.U., Tatabánya
- Italy (5):
  - For additional information regarding investigative sites for this trial, contact ITF Research Pharma S.L.U., Catania
  - For additional information regarding investigative sites for this trial, contact ITF Research Pharma S.L.U., Catanzaro
  - For additional information regarding investigative sites for this trial, contact ITF Research Pharma S.L.U., Modena
  - For additional information regarding investigative sites for this trial, contact ITF Research Pharma S.L.U., Pavia
  - For additional information regarding investigative sites for this trial, contact ITF Research Pharma S.L.U., Siena
- Spain (4):
  - For additional information regarding investigative sites for this trial, contact ITF Research Pharma S.L.U., Barcelona
  - For additional information regarding investigative sites for this trial, contact ITF Research Pharma S.L.U., Murcia
  - For additional information regarding investigative sites for this trial, contact ITF Research Pharma S.L.U., Santander
  - For additional information regarding investigative sites for this trial, contact ITF Research Pharma S.L.U., Valencia
- Sweden (3):
  - For additional information regarding investigative sites for this trial, contact ITF Research Pharma S.L.U., Huddinge
  - For additional information regarding investigative sites for this trial, contact ITF Research Pharma S.L.U., Kungsbacka
  - For additional information regarding investigative sites for this trial, contact ITF Research Pharma S.L.U., Stockholm

RESULTS

PARTICIPANT FLOW:
Groups:
- Estriol 0.005%: Subjects received 1 gram of Estriol 0.005% vaginal gel administered daily for Weeks 1-3. After 21 days of daily administration, treatment continued with twice-weekly administration up to Week 12
- Estriol 0.002%: Subjects received 1 gram of Estriol 0.002% vaginal gel administered daily for Weeks 1-3. After 21 days of daily administration, treatment continued with twice-weekly administration up to Week 12
- Estriol 0.0008%: Subjects received 1 gram of Estriol 0.0008% vaginal gel administered daily for Weeks 1-3. After 21 days of daily administration, treatment continued with twice-weekly administration up to Week 12
- Placebo: Subjects received 1 gram of matching placebo vaginal gel administered daily for Weeks 1-3. After 21 days of daily administration, treatment continued with twice-weekly administration up to Week 12
Period: Overall Study
Arm/Group | Estriol 0.005% | Estriol 0.002% | Estriol 0.0008% | Placebo
Started | 70 | 70 | 72 | 71
Completed | 66 | 67 | 65 | 63
Not Completed | 4 | 3 | 7 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Estriol 0.005% | Estriol 0.002% | Estriol 0.0008% | Placebo | Total
Number analyzed (Participants) | 70 | 70 | 72 | 71 | 283
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.5 (7.43) | 61.9 (6.87) | 62.2 (7.05) | 62.3 (7.24) | 62.0 (7.12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 70 | 70 | 72 | 71 | 283
  Male | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 70 | 70 | 71 | 71 | 282
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Week 12 in the Severity of Vaginal Dryness
Description: Percentage of Subjects with change from baseline to week 12 in the severity of vaginal dryness was reported. Severity was defined as: 0= Absent, 1= Mild, 2= Moderate, 3= Severe. A decrease in score compared to Baseline represented a positive outcome.
Time Frame: From baseline to week 12
Population: The ITT population defined as all randomized subjects. The number of subjects analyzed defined as number of subjects evaluable for this endpoint.
Measure: Count of Participants; unit: Participants
Arm/Group | Estriol 0.005% | Estriol 0.002% | Estriol 0.0008% | Placebo
Number analyzed (Participants) | 70 | 68 | 70 | 68
Participants
  Change from Baseline: -3 | 15 | 13 | 13 | 9
  Change from Baseline: -2 | 23 | 33 | 26 | 26
  Change from Baseline: -1 | 26 | 16 | 20 | 19
  Change from Baseline: 0 | 4 | 6 | 11 | 13
  Change from Baseline: 1 | 2 | 0 | 0 | 1
Statistical Analysis 1: Comparison: Estriol 0.005% vs Placebo; Test type: Superiority; p = 0.304, Wilcoxon rank-sum test — Hodges-Lehmann estimate (HLE) of median difference between treatments was calculated. Medians were not calculated per SAP as might cause confusion since the HLE of treatment difference is not identical to the difference between 2 treatment medians; Median Difference (Final Values) = 0, 95% CI 2-sided [-1 to 0] — Hodges-Lehmann estimate of location shift and corresponding asymptotic Confidence Interval
Statistical Analysis 2: Comparison: Estriol 0.002% vs Placebo; Test type: Superiority; p = 0.109, Wilcoxon rank-sum test — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0, 95% CI 2-sided [-1 to 0] — Hodges-Lehmann estimate of location shift and corresponding asymptotic Confidence Interval
Statistical Analysis 3: Comparison: Estriol 0.0008% vs Placebo; Test type: Superiority; p = 0.119, Wilcoxon rank-sum test — [p-value comment as in outcome 1, analysis 1]; Median Difference (Final Values) = 0, 95% CI 2-sided [0 to 0] — Hodges-Lehmann estimate of location shift and corresponding asymptotic Confidence Interval

2. Primary Outcome: Change From Baseline to Week 12 in Vaginal pH
Description: Change from Baseline to Week 12 in Vaginal pH was reported. A decrease in pH compare to Baseline represents a positive outcome.
Time Frame: Baseline to Week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: pH
Arm/Group | Estriol 0.005% | Estriol 0.002% | Estriol 0.0008% | Placebo
Number analyzed (Participants) | 70 | 68 | 70 | 69
pH | -1.03 (0.106) | -1.04 (0.108) | -0.95 (0.107) | -0.29 (0.108)
Statistical Analysis 1: Comparison: Estriol 0.005% vs Placebo; Test type: Superiority; p < 0.001, ANCOVA; LS Mean Difference = -0.74, 95% CI 2-sided [-1.031 to -0.444]
Statistical Analysis 2: Comparison: Estriol 0.002% vs Placebo; Test type: Superiority; p < 0.001, ANCOVA; LS Mean Difference = -0.75, 95% CI 2-sided [-1.051 to -0.458]
Statistical Analysis 3: Comparison: Estriol 0.0008% vs Placebo; Test type: Superiority; p < 0.001, ANCOVA; LS Mean Difference = -0.66, 95% CI 2-sided [-0.951 to -0.369]

3. Primary Outcome: Change From Baseline to Week 12 in the Proportion of Superficial Cells of the Vaginal Epithelium.
Description: Change from Baseline to week 12 in the proportion of superficial cells of the vaginal epithelium was reported.
Time Frame: Baseline to Week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: ratio
Arm/Group | Estriol 0.005% | Estriol 0.002% | Estriol 0.0008% | Placebo
Number analyzed (Participants) | 69 | 64 | 70 | 66
ratio | 0.24 (0.023) | 0.17 (0.024) | 0.19 (0.023) | 0.02 (0.024)
Statistical Analysis 1: Comparison: Estriol 0.005% vs Placebo; Test type: Superiority; p < 0.001, ANCOVA; LS Mean Difference = 0.21, 95% CI 2-sided [0.147 to 0.278]
Statistical Analysis 2: Comparison: Estriol 0.002% vs Placebo; Test type: Superiority; p < 0.001, ANCOVA; LS Mean Difference = 0.15, 95% CI 2-sided [0.078 to 0.213]
Statistical Analysis 3: Comparison: Estriol 0.0008% vs Placebo; Test type: Superiority; p < 0.001, ANCOVA; LS Mean Difference = 0.16, 95% CI 2-sided [0.097 to 0.226]

4. Primary Outcome: Change From Baseline to Week 12 in the Proportion of Parabasal Cells of the Vaginal Epithelium.
Description: Change from Baseline to Week 12 in the proportion of parabasal cells of the vaginal epithelium was reported. A decrease in proportion of parabasal cells compared to Baseline represents a positive outcome.
Time Frame: Baseline to Week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: ratio
Arm/Group | Estriol 0.005% | Estriol 0.002% | Estriol 0.0008% | Placebo
Number analyzed (Participants) | 69 | 64 | 70 | 66
ratio | -0.54 (0.036) | -0.51 (0.037) | -0.47 (0.036) | -0.04 (0.038)
Statistical Analysis 1: Comparison: Estriol 0.005% vs Placebo; Test type: Superiority; p < 0.001, ANCOVA; LS Mean Difference = -0.5, 95% CI 2-sided [-0.603 to -0.4]
Statistical Analysis 2: Comparison: Estriol 0.002% vs Placebo; Test type: Superiority; p < 0.001, ANCOVA; LS Mean Difference = -0.47, 95% CI 2-sided [-0.572 to -0.365]
Statistical Analysis 3: Comparison: Estriol 0.0008% vs Placebo; Test type: Superiority; p < 0.001, ANCOVA; LS Mean Difference = -0.43, 95% CI 2-sided [-0.531 to -0.331]

5. Secondary Outcome: Change From Baseline to Week 12 in the Severity of Dyspareunia
Description: Percentage of subjects with change from baseline to week 12 in the severity of dyspareunia was reported. Dyspareunia was only applicable in subjects who had experienced sexual activity with penetration since the previous study visit. Symptom scores at each visit: 0= Absent, 1= Mild, 2= Moderate, 3= Severe. A decrease in score compared to Baseline represented a positive outcome.
Time Frame: Baseline to Week 12
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Estriol 0.005% | Estriol 0.002% | Estriol 0.0008% | Placebo
Number analyzed (Participants) | 39 | 31 | 41 | 32
Participants
  Change from Baseline: -3 | 7 | 5 | 4 | 3
  Change from Baseline: -2 | 9 | 7 | 16 | 11
  Change from Baseline: -1 | 12 | 13 | 12 | 8
  Change from Baseline: 0 | 10 | 5 | 5 | 9
  Change from Baseline: 1 | 0 | 1 | 3 | 0
  Change from Baseline: 2 | 1 | 0 | 1 | 1
  Change from Baseline: 3 | 0 | 0 | 0 | 0
Statistical Analysis 1: Comparison: Estriol 0.005% vs Placebo; Test type: Superiority; p = 0.47, Wilcoxon rank-sum test — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0, 95% CI 2-sided [-1 to 0] — Hodges-Lehmann estimate of location shift and corresponding asymptotic Confidence Interval
Statistical Analysis 2: Comparison: Estriol 0.002% vs Placebo; Test type: Superiority; p = 0.448, Wilcoxon rank-sum test — [p-value comment as in outcome 1, analysis 1]; Median Difference (Final Values) = 0, 95% CI 2-sided [-1 to 0]; Hodges-Lehmann estimate of location shift and corresponding asymptotic Confidence Interval
Statistical Analysis 3: Comparison: Estriol 0.0008% vs Placebo; Test type: Superiority; p = 0.451, Wilcoxon rank-sum test — [p-value comment as in outcome 1, analysis 1]; Median Difference (Final Values) = 0, 95% CI 2-sided [-1 to 0] — Hodges-Lehmann estimate of location shift and corresponding asymptotic Confidence Interval

6. Secondary Outcome: Change From Baseline to Week 12 in the Severity of Pruritus or Itching
Description: Percentage of subjects with cvhange from Baseline to Week 12 in the severity of pruritus or itching was reported. Symptom scores at each visit: 0= Absent, 1= Mild, 2= Moderate, 3= Severe. A decrease in score compared to Baseline represented a positive outcome.
Time Frame: Baseline to Week 12
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Estriol 0.005% | Estriol 0.002% | Estriol 0.0008% | Placebo
Number analyzed (Participants) | 70 | 68 | 70 | 69
Participants
  Change from Baseline: -3 | 2 | 5 | 4 | 4
  Change from Baseline: -2 | 16 | 14 | 15 | 13
  Change from Baseline: -1 | 18 | 20 | 20 | 20
  Change from Baseline: 0 | 33 | 22 | 28 | 25
  Change from Baseline: 1 | 0 | 4 | 2 | 5
  Change from Baseline: 2 | 1 | 2 | 1 | 2
  Change from Baseline: 3 | 0 | 1 | 0 | 0
Statistical Analysis 1: Comparison: Estriol 0.005% vs Placebo; Test type: Superiority; p = 0.329, Wilcoxon rank-sum test — [p-value comment as in outcome 1, analysis 1]; Median Difference (Final Values) = 0, 95% CI 2-sided [0 to 0] — Hodges-Lehmann estimate of location shift and corresponding asymptotic Confidence Interval
Statistical Analysis 2: Comparison: Estriol 0.002% vs Placebo; Test type: Superiority; p = 0.348, Wilcoxon rank-sum test — [p-value comment as in outcome 1, analysis 1]; Median Difference (Final Values) = 0, 95% CI 2-sided [0 to 0] — Hodges-Lehmann estimate of location shift and corresponding asymptotic Confidence Interval
Statistical Analysis 3: Comparison: Estriol 0.0008% vs Placebo; Test type: Superiority; p = 0.266, Wilcoxon rank-sum test — [p-value comment as in outcome 1, analysis 1]; Median Difference (Final Values) = 0, 95% CI 2-sided [0 to 0] — Hodges-Lehmann estimate of location shift and corresponding asymptotic Confidence Interval

7. Secondary Outcome: Change From Baseline to Week 12 in the Severity of Burning
Description: Percentage of subjects with change from Baseline to Week 12 in the severity of burning was reported. Symptom scores at each visit: 0= Absent, 1= Mild, 2= Moderate, 3= Severe. A decrease in score compared to Baseline represented a positive outcome.
Time Frame: Baseline to Week 12
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Estriol 0.005% | Estriol 0.002% | Estriol 0.0008% | Placebo
Number analyzed (Participants) | 70 | 68 | 70 | 69
Participants
  Change from Baseline: -3 | 5 | 4 | 7 | 4
  Change from Baseline: -2 | 22 | 21 | 18 | 19
  Change from Baseline: -1 | 25 | 17 | 18 | 23
  Change from Baseline: 0 | 18 | 24 | 26 | 20
  Change from Baseline: 1 | 0 | 1 | 1 | 2
  Change from Baseline: 2 | 0 | 1 | 0 | 1
  Change from Baseline: 3 | 0 | 0 | 0 | 0
Statistical Analysis 1: Comparison: Estriol 0.005% vs Placebo; Test type: Superiority; p = 0.122, Wilcoxon rank-sum test — [p-value comment as in outcome 1, analysis 1]; Median Difference (Final Values) = 0, 95% CI 2-sided [0 to 0] — Hodges-Lehmann estimate of location shift and corresponding asymptotic Confidence Interval
Statistical Analysis 2: Comparison: Estriol 0.002% vs Placebo; Test type: Superiority; p = 0.188, Wilcoxon rank-sum test — [p-value comment as in outcome 1, analysis 1]; Median Difference (Final Values) = 0, 95% CI 2-sided [0 to 0] — Hodges-Lehmann estimate of location shift and corresponding asymptotic Confidence Interval
Statistical Analysis 3: Comparison: Estriol 0.0008% vs Placebo; Test type: Superiority; p = 0.222, Wilcoxon rank-sum test — [p-value comment as in outcome 1, analysis 1]; Median Difference (Final Values) = 0, 95% CI 2-sided [0 to 0] — Hodges-Lehmann estimate of location shift and corresponding asymptotic Confidence Interval

8. Secondary Outcome: Change From Baseline to Week 12 in the Severity of Dysuria
Description: Percentage of subjects with change from Baseline to Week 12 in the severity of dysuria was reported. Symptom scores at each visit: 0= Absent, 1= Mild, 2= Moderate, 3= Severe. A decrease in score compared to baseline represented a positive putcome.
Time Frame: Baseline to Week 12
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Estriol 0.005% | Estriol 0.002% | Estriol 0.0008% | Placebo
Number analyzed (Participants) | 70 | 68 | 70 | 69
Participants
  Change from Baseline: -3 | 0 | 1 | 1 | 1
  Change from Baseline: -2 | 8 | 8 | 5 | 5
  Change from Baseline: -1 | 18 | 19 | 17 | 15
  Change from Baseline: 0 | 43 | 39 | 40 | 44
  Change from Baseline: 1 | 1 | 1 | 7 | 0
  Change from Baseline: 2 | 0 | 0 | 0 | 2
  Change from Baseline: 3 | 0 | 0 | 0 | 2
Statistical Analysis 1: Comparison: Estriol 0.005% vs Placebo; Test type: Superiority; p = 0.393, Wilcoxon rank-sum test — [p-value comment as in outcome 1, analysis 1]; Median Difference (Final Values) = 0, 95% CI 2-sided [0 to 0] — Hodges-Lehmann estimate of location shift and corresponding asymptotic Confidence Interval
Statistical Analysis 2: Comparison: Estriol 0.002% vs Placebo; Test type: Superiority; p = 0.221, Wilcoxon rank-sum test — [p-value comment as in outcome 1, analysis 1]; Median Difference (Final Values) = 0, 95% CI 2-sided [0 to 0] — Hodges-Lehmann estimate of location shift and corresponding asymptotic Confidence Interval
Statistical Analysis 3: Comparison: Estriol 0.0008% vs Placebo; Test type: Superiority; p = 0.432, Wilcoxon rank-sum test — [p-value comment as in outcome 1, analysis 1]; Median Difference (Final Values) = 0, 95% CI 2-sided [0 to 0] — Hodges-Lehmann estimate of location shift and corresponding asymptotic Confidence Interval

9. Secondary Outcome: Change From Baseline to Week 12 in the Global Symptom Score 1
Description: Global Symptom Score 1 was defined as the sum of all 5 individual symptom scores at a given visit, and was calculated only when all 5 symptom scores had a response available. the Global Symptom Score 1 ranged at Screening/Baseline between 2 (at least moderate vaginal dryness -per inclusion criteria) to 15 (all 5 studied symptoms severe in intensity). At Week 12/ET visit, the Global Symptom Score ranged between 0 (no symptoms) and 15 (all symptoms severe in intensity). A decrease in score compared to Baseline represented a positive outcome.
Time Frame: Baseline to Week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Estriol 0.005% | Estriol 0.002% | Estriol 0.0008% | Placebo
Number analyzed (Participants) | 39 | 31 | 41 | 31
units on a scale | -4.30 (0.425) | -4.78 (0.478) | -4.51 (0.412) | -4.54 (0.467)
Statistical Analysis 1: Comparison: Estriol 0.005% vs Placebo; Test type: Superiority; p = 0.65, ANCOVA; LS Mean Difference = 0.24, 95% CI 2-sided [-1 to 1.487]
Statistical Analysis 2: Comparison: Estriol 0.002% vs Placebo; Test type: Superiority; p = 0.361, ANCOVA; LS Mean Difference = -0.24, 95% CI 2-sided [-1.568 to 1.09]
Statistical Analysis 3: Comparison: Estriol 0.0008% vs Placebo; Test type: Superiority; p = 0.522, ANCOVA; LS Mean Difference = 0.03, 95% CI 2-sided [-1.188 to 1.257]

10. Secondary Outcome: Change From Baseline to Week 12 in the Global Symptom Score 2
Description: Change from Baseline to Week 12 in the Global Symptom Score 2 was reported. Global Symptom Score 2 was defined as the sum of all 4 individual symptoms excluding dyspareunia (vaginal dryness, pruritus or itching, burning, and dysuria) for each subject at each time point: Screening/Baseline, Week 3 and Week 12/ET., and was calculated only when all 4 symptom scores had a response available. The maximum score possible to be obtained at a visit with the Global Symptom Score 2 was 12 (all symptoms severe in intensity). A decrease in score compared to baseline represented a positive outcome.
Time Frame: Baseline to Week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Estriol 0.005% | Estriol 0.002% | Estriol 0.0008% | Placebo
Number analyzed (Participants) | 70 | 68 | 70 | 68
units on a scale | -3.83 (0.231) | -3.78 (0.234) | -3.74 (0.233) | -3.27 (0.237)
Statistical Analysis 1: Comparison: Estriol 0.005% vs Placebo; Test type: Superiority; p = 0.043, ANCOVA; LS Mean Difference = -0.56, 95% CI 2-sided [-1.204 to 0.079]
Statistical Analysis 2: Comparison: Estriol 0.002% vs Placebo; Test type: Superiority; p = 0.061, ANCOVA; LS Mean Difference = -0.51, 95% CI 2-sided [-1.158 to 0.137]
Statistical Analysis 3: Comparison: Estriol 0.0008% vs Placebo; Test type: Superiority; p = 0.071, ANCOVA; LS Mean Difference = -0.48, 95% CI 2-sided [-1.111 to 0.16]

11. Secondary Outcome: Change From Baseline to Week 12 in the Severity of Pallor.
Description: Percentage of subjects with change from Baseline to Week 12 in the severity of pallor was reported. Sign scores at each visit: 0= Absent, 1= Mild, 2= Moderate, 3= Severe. A decrease in score compared to baseline represented a positive putcome.
Time Frame: Baseline to Week 12
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Estriol 0.005% | Estriol 0.002% | Estriol 0.0008% | Placebo
Number analyzed (Participants) | 70 | 68 | 70 | 69
Participants
  Change from Baseline: -3 | 3 | 5 | 1 | 1
  Change from Baseline: -2 | 17 | 16 | 25 | 15
  Change from Baseline: -1 | 31 | 31 | 25 | 18
  Change from Baseline: 0 | 16 | 16 | 17 | 31
  Change from Baseline: 1 | 3 | 0 | 2 | 4
  Change from Baseline: 2 | 0 | 0 | 0 | 0
  Change from Baseline: 3 | 0 | 0 | 0 | 0
Statistical Analysis 1: Comparison: Estriol 0.005% vs Placebo; Test type: Superiority; p = 0.012, Wilcoxon rank-sum test — [p-value comment as in outcome 1, analysis 1]; Median Difference (Final Values) = 0, 95% CI 2-sided [-1 to 0] — Hodges-Lehmann estimate of location shift and corresponding asymptotic Confidence Interval
Statistical Analysis 2: Comparison: Estriol 0.002% vs Placebo; Test type: Superiority; p = 0.007, Wilcoxon rank-sum test — [p-value comment as in outcome 1, analysis 1]; Median Difference (Final Values) = 0, 95% CI 2-sided [-1 to 0] — Hodges-Lehmann estimate of location shift and corresponding asymptotic Confidence Interval
Statistical Analysis 3: Comparison: Estriol 0.0008% vs Placebo; Test type: Superiority; p < 0.001, Wilcoxon rank-sum test — [p-value comment as in outcome 1, analysis 1]; Median Difference (Final Values) = 0, 95% CI 2-sided [-1 to 0] — Hodges-Lehmann estimate of location shift and corresponding asymptotic Confidence Interval

12. Secondary Outcome: Change From Baseline to Week 12 in the Severity of Friability
Description: Percentage of subjects with change from Baseline to Week 12 in the severity of friability was reported. Sign scores at each visit: 0= Absent, 1= Mild, 2= Moderate, 3= Severe. A decrease in score compared to baseline represented a positive outcome.
Time Frame: Baseline to Week 12
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Estriol 0.005% | Estriol 0.002% | Estriol 0.0008% | Placebo
Number analyzed (Participants) | 70 | 68 | 70 | 69
Participants
  Change from Baseline: -3 | 2 | 2 | 2 | 3
  Change from Baseline: -2 | 19 | 21 | 18 | 19
  Change from Baseline: -1 | 26 | 22 | 31 | 20
  Change from Baseline: 0 | 21 | 22 | 16 | 24
  Change from Baseline: 1 | 1 | 0 | 3 | 3
  Change from Baseline: 2 | 1 | 1 | 0 | 0
  Change from Baseline: 3 | 0 | 0 | 0 | 0
Statistical Analysis 1: Comparison: Estriol 0.005% vs Placebo; Test type: Superiority; p = 0.438, Wilcoxon rank-sum test — [p-value comment as in outcome 1, analysis 1]; Median Difference (Final Values) = 0, 95% CI 2-sided [0 to 0] — Hodges-Lehmann estimate of location shift and corresponding asymptotic Confidence Interval
Statistical Analysis 2: Comparison: Estriol 0.002% vs Placebo; Test type: Superiority; p = 0.388, Wilcoxon rank-sum test — [p-value comment as in outcome 1, analysis 1]; Median Difference (Final Values) = 0, 95% CI 2-sided [0 to 0] — Hodges-Lehmann estimate of location shift and corresponding asymptotic Confidence Interval
Statistical Analysis 3: Comparison: Estriol 0.0008% vs Placebo; Test type: Superiority; p = 0.259, Wilcoxon rank-sum test — [p-value comment as in outcome 1, analysis 1]; Median Difference (Final Values) = 0, 95% CI 2-sided [0 to 0] — Hodges-Lehmann estimate of location shift and corresponding asymptotic Confidence Interval

13. Secondary Outcome: Change From Baseline to Week 12 in the Severity of Thinning or Flattening of Folds
Description: Percentage of subjects with change from Baseline to Week 12 in the severity of thinning or flattening of folds was reported. Sign scores at each visit: 0= Absent, 1= Mild, 2= Moderate, 3= Severe. A decrease in score compared to baseline represented a positive outcome.
Time Frame: Baseline to Week 12
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Estriol 0.005% | Estriol 0.002% | Estriol 0.0008% | Placebo
Number analyzed (Participants) | 70 | 68 | 70 | 69
Participants
  Change from Baseline: -3 | 4 | 1 | 1 | 1
  Change from Baseline: -2 | 18 | 18 | 23 | 6
  Change from Baseline: -1 | 29 | 33 | 24 | 31
  Change from Baseline: 0 | 17 | 14 | 19 | 26
  Change from Baseline: 1 | 2 | 2 | 3 | 5
  Change from Baseline: 2 | 0 | 0 | 0 | 0
  Change from Baseline: 3 | 0 | 0 | 0 | 0
Statistical Analysis 1: Comparison: Estriol 0.005% vs Placebo; Test type: Superiority; p = 0.022, Wilcoxon rank-sum test — [p-value comment as in outcome 1, analysis 1]; Median Difference (Final Values) = 0, 95% CI 2-sided [-1 to 0] — Hodges-Lehmann estimate of location shift and corresponding asymptotic Confidence Interval
Statistical Analysis 2: Comparison: Estriol 0.002% vs Placebo; Test type: Superiority; p = 0.02, Wilcoxon rank-sum test — [p-value comment as in outcome 1, analysis 1]; Median Difference (Final Values) = 0, 95% CI 2-sided [-1 to 0] — Hodges-Lehmann estimate of location shift and corresponding asymptotic Confidence Interval
Statistical Analysis 3: Comparison: Estriol 0.0008% vs Placebo; Test type: Superiority; p = 0.003, Wilcoxon rank-sum test — [p-value comment as in outcome 1, analysis 1]; Median Difference (Final Values) = 0, 95% CI 2-sided [-1 to 0] — Hodges-Lehmann estimate of location shift and corresponding asymptotic Confidence Interval

14. Secondary Outcome: Change From Baseline to Week 12 in the Severity of Petechiae
Description: Percentage of subjects with change from Baseline to Week 12 in the severity of presence of petechiae was reported. Sign scores at each visit: 0= Absent, 1= Mild, 2= Moderate, 3= Severe. A decrease in score compared to baseline represented a positive outcome.
Time Frame: Baseline to Week 12
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Estriol 0.005% | Estriol 0.002% | Estriol 0.0008% | Placebo
Number analyzed (Participants) | 70 | 68 | 70 | 69
Participants
  Change from Baseline: -3 | 2 | 1 | 0 | 2
  Change from Baseline: -2 | 10 | 5 | 7 | 2
  Change from Baseline: -1 | 26 | 23 | 23 | 13
  Change from Baseline: 0 | 29 | 35 | 35 | 49
  Change from Baseline: 1 | 3 | 4 | 5 | 3
  Change from Baseline: 2 | 0 | 0 | 0 | 0
  Change from Baseline: 3 | 0 | 0 | 0 | 0
Statistical Analysis 1: Comparison: Estriol 0.005% vs Placebo; Test type: Superiority; p = 0.002, Wilcoxon rank-sum test — [p-value comment as in outcome 1, analysis 1]; Median Difference (Final Values) = 0, 95% CI 2-sided [-1 to 0] — Hodges-Lehmann estimate of location shift and corresponding asymptotic Confidence Interval
Statistical Analysis 2: Comparison: Estriol 0.002% vs Placebo; Test type: Superiority; p = 0.331, Wilcoxon rank-sum test — [p-value comment as in outcome 1, analysis 1]; Median Difference (Final Values) = 0, 95% CI 2-sided [0 to 0] — Hodges-Lehmann estimate of location shift and corresponding asymptotic Confidence Interval
Statistical Analysis 3: Comparison: Estriol 0.0008% vs Placebo; Test type: Superiority; p = 0.043, Wilcoxon rank-sum test — [p-value comment as in outcome 1, analysis 1]; Median Difference (Final Values) = 0, 95% CI 2-sided [0 to 0] — Hodges-Lehmann estimate of location shift and corresponding asymptotic Confidence Interval

15. Secondary Outcome: Change From Baseline to Week 12 in the Severity of Dry Mucosa
Description: Percentage of subjects with change from Baseline to Week 12 in the severity of dry mucosa was reported. Sign scores at each visit: 0= Absent, 1= Mild, 2= Moderate, 3= Severe. A decrease in score compared to baseline represented a positive outcome.
Time Frame: Baseline to Week 12
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Estriol 0.005% | Estriol 0.002% | Estriol 0.0008% | Placebo
Number analyzed (Participants) | 70 | 68 | 70 | 69
Participants
  Change from Baseline: -3 | 8 | 13 | 14 | 9
  Change from Baseline: -2 | 39 | 29 | 26 | 19
  Change from Baseline: -1 | 17 | 20 | 23 | 19
  Change from Baseline: 0 | 5 | 6 | 6 | 19
  Change from Baseline: 1 | 1 | 0 | 1 | 3
  Change from Baseline: 2 | 0 | 0 | 0 | 0
  Change from Baseline: 3 | 0 | 0 | 0 | 0
Statistical Analysis 1: Comparison: Estriol 0.005% vs Placebo; Test type: Superiority; p = 0.022, Wilcoxon rank-sum test — [p-value comment as in outcome 1, analysis 1]; Median Difference (Final Values) = -1, 95% CI 2-sided [-1 to 0] — Hodges-Lehmann estimate of location shift and corresponding asymptotic Confidence Interval
Statistical Analysis 2: Comparison: Estriol 0.002% vs Placebo; Test type: Superiority; p = 0.032, Wilcoxon rank-sum test — [p-value comment as in outcome 1, analysis 1]; Median Difference (Final Values) = -1, 95% CI 2-sided [-1 to 0] — Hodges-Lehmann estimate of location shift and corresponding asymptotic Confidence Interval
Statistical Analysis 3: Comparison: Estriol 0.0008% vs Placebo; Test type: Superiority; p = 0.001, Wilcoxon rank-sum test — [p-value comment as in outcome 1, analysis 1]; Median Difference (Final Values) = -1, 95% CI 2-sided [-1 to 0] — Hodges-Lehmann estimate of location shift and corresponding asymptotic Confidence Interval

16. Secondary Outcome: Change From Baseline to Week 3 in the Severity of Vaginal Dryness
Description: Percentage of subjects with change from Baseline to Week 3 in the severity of vaginal dryness was reported. Severity was defined as: 0= Absent, 1= Mild, 2= Moderate, 3= Severe. A decrease in score compared to baseline represented a positive outcome.
Time Frame: Baseline to Week 3
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Estriol 0.005% | Estriol 0.002% | Estriol 0.0008% | Placebo
Number analyzed (Participants) | 68 | 66 | 68 | 68
Participants
  Change from Baseline: -3 | 6 | 8 | 8 | 3
  Change from Baseline: -2 | 23 | 13 | 22 | 26
  Change from Baseline: -1 | 28 | 33 | 26 | 26
  Change from Baseline: 0 | 8 | 12 | 11 | 11
  Change from Baseline: 1 | 3 | 0 | 1 | 2
Statistical Analysis 1: Comparison: Estriol 0.005% vs Placebo; Test type: Superiority; p = 0.176, Wilcoxon rank-sum test — [p-value comment as in outcome 1, analysis 1]; Median Difference (Final Values) = 0, 95% CI 2-sided [0 to 0] — Hodges-Lehmann estimate of location shift and corresponding asymptotic Confidence Interval
Statistical Analysis 2: Comparison: Estriol 0.002% vs Placebo; Test type: Superiority; p = 0.358, Wilcoxon rank-sum test — [p-value comment as in outcome 1, analysis 1]; Median Difference (Final Values) = 0, 95% CI 2-sided [0 to 0] — Hodges-Lehmann estimate of location shift and corresponding asymptotic Confidence Interval
Statistical Analysis 3: Comparison: Estriol 0.0008% vs Placebo; Test type: Superiority; p = 0.21, Wilcoxon rank-sum test — [p-value comment as in outcome 1, analysis 1]; Median Difference (Final Values) = 0, 95% CI 2-sided [0 to 0] — Hodges-Lehmann estimate of location shift and corresponding asymptotic Confidence Interval

17. Secondary Outcome: Change From Baseline to Week 3 in the Severity of Dyspareunia
Description: Percentage of subjects with change from Baseline to Week 3 in severity of dyspareunia was reported. Dyspareunia was only applicable in subjects who had experienced sexual activity with penetration since the previous study visit. Symptom scores at each visit: 0= Absent, 1= Mild, 2= Moderate, 3= Severe. A decrease in score compared to baseline represented a positive outcome.
Time Frame: From baseline to week 3
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Estriol 0.005% | Estriol 0.002% | Estriol 0.0008% | Placebo
Number analyzed (Participants) | 33 | 29 | 37 | 27
Participants
  Change from Baseline: -3 | 1 | 3 | 4 | 2
  Change from Baseline: -2 | 7 | 4 | 10 | 7
  Change from Baseline: -1 | 11 | 11 | 14 | 10
  Change from Baseline: 0 | 13 | 6 | 8 | 7
  Change from Baseline: 1 | 0 | 4 | 0 | 1
  Change from Baseline: 2 | 1 | 1 | 1 | 0
  Change from Baseline: 3 | 0 | 0 | 0 | 0
Statistical Analysis 1: Comparison: Estriol 0.005% vs Placebo; Test type: Superiority; p = 0.106, Wilcoxon rank-sum test — [p-value comment as in outcome 1, analysis 1]; Median Difference (Final Values) = 0, 95% CI 2-sided [0 to 1] — Hodges-Lehmann estimate of location shift and corresponding asymptotic Confidence Interval
Statistical Analysis 2: Comparison: Estriol 0.002% vs Placebo; Test type: Superiority; p = 0.229, Wilcoxon rank-sum test — [p-value comment as in outcome 1, analysis 1]; Median Difference (Final Values) = 0, 95% CI 2-sided [0 to 1] — Hodges-Lehmann estimate of location shift and corresponding asymptotic Confidence Interval
Statistical Analysis 3: Comparison: Estriol 0.0008% vs Placebo; Test type: Superiority; p = 0.345, Wilcoxon rank-sum test — [p-value comment as in outcome 1, analysis 1]; Median Difference (Final Values) = 0, 95% CI 2-sided [-1 to 0] — Hodges-Lehmann estimate of location shift and corresponding asymptotic Confidence Interval

18. Secondary Outcome: Change From Baseline to Week 3 in the Severity of Pruritus or Itching
Description: Percentage of subjects with change from Baseline to Week 3 in the severity of pruritus or itching was reported. Symptom scores at each visit: 0= Absent, 1= Mild, 2= Moderate, 3= Severe. A decrease in score compared to baseline represented a positive outcome.
Time Frame: Baseline to Week 3
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Estriol 0.005% | Estriol 0.002% | Estriol 0.0008% | Placebo
Number analyzed (Participants) | 68 | 67 | 68 | 68
Participants
  Change from Baseline: -3 | 1 | 4 | 2 | 1
  Change from Baseline: -2 | 10 | 10 | 7 | 10
  Change from Baseline: -1 | 15 | 19 | 30 | 24
  Change from Baseline: 0 | 35 | 27 | 27 | 30
  Change from Baseline: 1 | 5 | 2 | 2 | 0
  Change from Baseline: 2 | 2 | 4 | 0 | 3
  Change from Baseline: 3 | 0 | 1 | 0 | 0
Statistical Analysis 1: Comparison: Estriol 0.005% vs Placebo; Test type: Superiority; p = 0.026, Wilcoxon rank-sum test — [p-value comment as in outcome 1, analysis 1]; Median Difference (Final Values) = 0, 95% CI 2-sided [0 to 0] — Hodges-Lehmann estimate of location shift and corresponding asymptotic Confidence Interval
Statistical Analysis 2: Comparison: Estriol 0.002% vs Placebo; Test type: Superiority; p = 0.424, Wilcoxon rank-sum test — [p-value comment as in outcome 1, analysis 1]; Median Difference (Final Values) = 0, 95% CI 2-sided [0 to 0] — Hodges-Lehmann estimate of location shift and corresponding asymptotic Confidence Interval
Statistical Analysis 3: Comparison: Estriol 0.0008% vs Placebo; Test type: Superiority; p = 0.414, Wilcoxon rank-sum test — [p-value comment as in outcome 1, analysis 1]; Median Difference (Final Values) = 0, 95% CI 2-sided [0 to 0] — Hodges-Lehmann estimate of location shift and corresponding asymptotic Confidence Interval

19. Secondary Outcome: Change From Baseline to Week 3 in the Severity of Burning
Description: Percentage of subjects with change from Baseline to Week 3 in severity of burning was reported. Symptom scores at each visit: 0= Absent, 1= Mild, 2= Moderate, 3= Severe. A decrease in score compared to baseline represented a positive outcome.
Time Frame: Baseline to Week 3
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Estriol 0.005% | Estriol 0.002% | Estriol 0.0008% | Placebo
Number analyzed (Participants) | 68 | 67 | 68 | 68
Participants
  Change from Baseline: -3 | 3 | 2 | 4 | 0
  Change from Baseline: -2 | 11 | 17 | 14 | 16
  Change from Baseline: -1 | 27 | 18 | 20 | 21
  Change from Baseline: 0 | 27 | 28 | 29 | 28
  Change from Baseline: 1 | 0 | 1 | 1 | 2
  Change from Baseline: 2 | 0 | 1 | 0 | 1
  Change from Baseline: 3 | 0 | 0 | 0 | 0
Statistical Analysis 1: Comparison: Estriol 0.005% vs Placebo; Test type: Superiority; p = 0.36, Wilcoxon rank-sum test — [p-value comment as in outcome 1, analysis 1]; Median Difference (Final Values) = 0, 95% CI 2-sided [0 to 0] — Hodges-Lehmann estimate of location shift and corresponding asymptotic Confidence Interval
Statistical Analysis 2: Comparison: Estriol 0.002% vs Placebo; Test type: Superiority; p = 0.12, Wilcoxon rank-sum test — [p-value comment as in outcome 1, analysis 1]; Median Difference (Final Values) = 0, 95% CI 2-sided [0 to 0] — Hodges-Lehmann estimate of location shift and corresponding asymptotic Confidence Interval
Statistical Analysis 3: Comparison: Estriol 0.0008% vs Placebo; Test type: Superiority; p = 0.266, Wilcoxon rank-sum test — [p-value comment as in outcome 1, analysis 1]; Median Difference (Final Values) = 0, 95% CI 2-sided [0 to 0] — Hodges-Lehmann estimate of location shift and corresponding asymptotic Confidence Interval

20. Secondary Outcome: Change From Baseline to Week 3 in the Severity of Dysuria
Description: Percentage of subjects with change from Baseline to Week 3 in severity of dysuria was reported. Symptom scores at each visit: 0= Absent, 1= Mild, 2= Moderate, 3= Severe. A decrease in score compared to baseline represented a positive outcome.
Time Frame: Baseline to Week 3
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Estriol 0.005% | Estriol 0.002% | Estriol 0.0008% | Placebo
Number analyzed (Participants) | 68 | 67 | 68 | 68
Participants
  Change from Baseline: -3 | 0 | 0 | 1 | 0
  Change from Baseline: -2 | 5 | 8 | 3 | 6
  Change from Baseline: -1 | 14 | 16 | 14 | 9
  Change from Baseline: 0 | 46 | 39 | 48 | 48
  Change from Baseline: 1 | 3 | 3 | 2 | 3
  Change from Baseline: 2 | 0 | 0 | 0 | 0
  Change from Baseline: 3 | 0 | 1 | 0 | 2
Statistical Analysis 1: Comparison: Estriol 0.005% vs Placebo; Test type: Superiority; p = 0.47, Wilcoxon rank-sum test — [p-value comment as in outcome 1, analysis 1]; Median Difference (Final Values) = 0, 95% CI 2-sided [0 to 0] — Hodges-Lehmann estimate of location shift and corresponding asymptotic Confidence Interval
Statistical Analysis 2: Comparison: Estriol 0.002% vs Placebo; Test type: Superiority; p = 0.137, Wilcoxon rank-sum test — [p-value comment as in outcome 1, analysis 1]; Median Difference (Final Values) = 0, 95% CI 2-sided [0 to 0] — Hodges-Lehmann estimate of location shift and corresponding asymptotic Confidence Interval
Statistical Analysis 3: Comparison: Estriol 0.0008% vs Placebo; Test type: Superiority; p = 0.133, Wilcoxon rank-sum test — [p-value comment as in outcome 1, analysis 1]; Median Difference (Final Values) = 0, 95% CI 2-sided [0 to 0] — Hodges-Lehmann estimate of location shift and corresponding asymptotic Confidence Interval

21. Secondary Outcome: Change From Baseline to Week 3 in the Global Symptom Score 1
Description: Global Symptom Score 1 was defined as the sum of all 5 individual symptom scores at a given visit, and was calculated only when all 5 symptom scores had a response available. the Global Symptom Score 1 ranged at Screening/Baseline between 2 (at least moderate vaginal dryness -per inclusion criteria) to 15 (all 5 studied symptoms severe in intensity). At Week 3 visit, the Global Symptom Score ranged between 0 (no symptoms) and 15 (all symptoms severe in intensity). A decrease in score compared to Baseline represented a positive outcome.
Time Frame: Baseline to Week 3
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Estriol 0.005% | Estriol 0.002% | Estriol 0.0008% | Placebo
Number analyzed (Participants) | 33 | 29 | 37 | 27
units on a scale | -2.99 (0.483) | -2.86 (0.520) | -4.37 (0.454) | -3.73 (0.527)
Statistical Analysis 1: Comparison: Estriol 0.005% vs Placebo; Test type: Superiority; p = 0.85, ANCOVA; LS Mean Difference = 0.74, 95% CI 2-sided [-0.669 to 2.153]
Statistical Analysis 2: Comparison: Estriol 0.002% vs Placebo; Test type: Superiority; p = 0.877, ANCOVA; LS Mean Difference = 0.87, 95% CI 2-sided [-0.611 to 2.361]
Statistical Analysis 3: Comparison: Estriol 0.0008% vs Placebo; Test type: Superiority; p = 0.178, ANCOVA; LS Mean Difference = -0.64, 95% CI 2-sided [-2.009 to 0.728]

22. Secondary Outcome: Change From Baseline to Week 3 in the Global Symptom Score 2
Description: Change from Baseline to Week 3 in the Global Symptom Score 2 was reported. Global Symptom Score 2 was defined as the sum of all 4 individual symptoms excluding dyspareunia (vaginal dryness, pruritus or itching, burning, and dysuria) for each subject at each time point: Screening/Baseline, Week 3 and Week 12/ET., and was calculated only when all 4 symptom scores had a response available. The maximum score possible to be obtained at a visit with the Global Symptom Score 2 was 12 (all symptoms severe in intensity). A decrease in score compared to baseline represented a positive outcome.
Time Frame: Baseline to Week 3
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Estriol 0.005% | Estriol 0.002% | Estriol 0.0008% | Placebo
Number analyzed (Participants) | 68 | 66 | 68 | 68
units on a scale | -2.76 (0.251) | -2.82 (0.254) | -3.20 (0.253) | -2.60 (0.255)
Statistical Analysis 1: Comparison: Estriol 0.005% vs Placebo; Test type: Superiority; p = 0.323, ANCOVA; LS Mean Difference = -0.16, 95% CI 2-sided [-0.854 to 0.531]
Statistical Analysis 2: Comparison: Estriol 0.002% vs Placebo; Test type: Superiority; p = 0.272, ANCOVA; LS Mean Difference = -0.22, 95% CI 2-sided [-0.917 to 0.484]
Statistical Analysis 3: Comparison: Estriol 0.0008% vs Placebo; Test type: Superiority; p = 0.043, ANCOVA; LS Mean Difference = -0.6, 95% CI 2-sided [-1.29 to 0.084]

23. Secondary Outcome: Change From Baseline to Week 3 in the Severity of Pallor
Description: Percentage of subjects with change from Baseline to Week 3 in severity of pallor was reported. Sign scores at each visit: 0= Absent, 1= Mild, 2= Moderate, 3= Severe. A decrease in score compared to baseline represented a positive outcome.
Time Frame: Baseline to Week 3
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Estriol 0.005% | Estriol 0.002% | Estriol 0.0008% | Placebo
Number analyzed (Participants) | 68 | 67 | 68 | 68
Participants
  Change from Baseline: -3 | 3 | 2 | 1 | 0
  Change from Baseline: -2 | 14 | 14 | 14 | 6
  Change from Baseline: -1 | 19 | 20 | 24 | 19
  Change from Baseline: 0 | 31 | 30 | 29 | 38
  Change from Baseline: 1 | 1 | 1 | 0 | 5
  Change from Baseline: 2 | 0 | 0 | 0 | 0
  Change from Baseline: 3 | 0 | 0 | 0 | 0
Statistical Analysis 1: Comparison: Estriol 0.005% vs Placebo; Test type: Superiority; p = 0.009, Wilcoxon rank-sum test — [p-value comment as in outcome 1, analysis 1]; Median Difference (Final Values) = 0, 95% CI 2-sided [-1 to 0] — Hodges-Lehmann estimate of location shift and corresponding asymptotic Confidence Interval
Statistical Analysis 2: Comparison: Estriol 0.002% vs Placebo; Test type: Superiority; p = 0.025, Wilcoxon rank-sum test — [p-value comment as in outcome 1, analysis 1]; Median Difference (Final Values) = 0, 95% CI 2-sided [-1 to 0] — Hodges-Lehmann estimate of location shift and corresponding asymptotic Confidence Interval
Statistical Analysis 3: Comparison: Estriol 0.0008% vs Placebo; Test type: Superiority; p < 0.001, Wilcoxon rank-sum test — [p-value comment as in outcome 1, analysis 1]; Median Difference (Final Values) = 0, 95% CI 2-sided [-1 to 0] — Hodges-Lehmann estimate of location shift and corresponding asymptotic Confidence Interval

24. Secondary Outcome: Change From Baseline to Week 3 in the Severity of Friability
Description: Percentage of subjects with change from Baseline to Week 3 in severity of friability was reported. Sign scores at each visit: 0= Absent, 1= Mild, 2= Moderate, 3= Severe. A decrease in score compared to baseline represented a positive outcome.
Time Frame: Baseline to Week 3
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Estriol 0.005% | Estriol 0.002% | Estriol 0.0008% | Placebo
Number analyzed (Participants) | 68 | 67 | 68 | 68
Participants
  Change from Baseline: -3 | 2 | 2 | 1 | 0
  Change from Baseline: -2 | 14 | 11 | 13 | 9
  Change from Baseline: -1 | 29 | 25 | 25 | 24
  Change from Baseline: 0 | 22 | 25 | 27 | 32
  Change from Baseline: 1 | 1 | 3 | 2 | 3
  Change from Baseline: 2 | 0 | 1 | 0 | 0
  Change from Baseline: 3 | 0 | 0 | 0 | 0
Statistical Analysis 1: Comparison: Estriol 0.005% vs Placebo; Test type: Superiority; p = 0.04, Wilcoxon rank-sum test — [p-value comment as in outcome 1, analysis 1]; Median Difference (Final Values) = 0, 95% CI 2-sided [-1 to 0] — Hodges-Lehmann estimate of location shift and corresponding asymptotic Confidence Interval
Statistical Analysis 2: Comparison: Estriol 0.002% vs Placebo; Test type: Superiority; p = 0.259, Wilcoxon rank-sum test — [p-value comment as in outcome 1, analysis 1]; Median Difference (Final Values) = 0, 95% CI 2-sided [0 to 0] — Hodges-Lehmann estimate of location shift and corresponding asymptotic Confidence Interval
Statistical Analysis 3: Comparison: Estriol 0.0008% vs Placebo; Test type: Superiority; p = 0.104, Wilcoxon rank-sum test — [p-value comment as in outcome 1, analysis 1]; Median Difference (Final Values) = 0, 95% CI 2-sided [0 to 0] — Hodges-Lehmann estimate of location shift and corresponding asymptotic Confidence Interval

25. Secondary Outcome: Change From Baseline to Week 3 in the Severity of Thinning or Flattening of Folds
Description: Percentage of subjects with change from Baseline to Week 3 in severity of thinning or flattening of folds was reported. Sign scores at each visit: 0= Absent, 1= Mild, 2= Moderate, 3= Severe. A decrease in score compared to baseline represented a positive outcome.
Time Frame: Baseline to Week 3
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Estriol 0.005% | Estriol 0.002% | Estriol 0.0008% | Placebo
Number analyzed (Participants) | 68 | 67 | 68 | 68
Participants
  Change from Baseline: -3 | 1 | 1 | 0 | 0
  Change from Baseline: -2 | 12 | 9 | 10 | 5
  Change from Baseline: -1 | 32 | 35 | 31 | 16
  Change from Baseline: 0 | 20 | 21 | 26 | 43
  Change from Baseline: 1 | 3 | 1 | 1 | 4
  Change from Baseline: 2 | 0 | 0 | 0 | 0
  Change from Baseline: 3 | 0 | 0 | 0 | 0
Statistical Analysis 1: Comparison: Estriol 0.005% vs Placebo; Test type: Superiority; p < 0.001, Wilcoxon rank-sum test — [p-value comment as in outcome 1, analysis 1]; Median Difference (Final Values) = -1, 95% CI 2-sided [-1 to 0] — Hodges-Lehmann estimate of location shift and corresponding asymptotic Confidence Interval
Statistical Analysis 2: Comparison: Estriol 0.002% vs Placebo; Test type: Superiority; p < 0.001, Wilcoxon rank-sum test — [p-value comment as in outcome 1, analysis 1]; Median Difference (Final Values) = -1, 95% CI 2-sided [-1 to 0] — Hodges-Lehmann estimate of location shift and corresponding asymptotic Confidence Interval
Statistical Analysis 3: Comparison: Estriol 0.0008% vs Placebo; Test type: Superiority; p < 0.001, Wilcoxon rank-sum test — [p-value comment as in outcome 1, analysis 1]; Median Difference (Final Values) = 0, 95% CI 2-sided [-1 to 0] — Hodges-Lehmann estimate of location shift and corresponding asymptotic Confidence Interval

26. Secondary Outcome: Change From Baseline to Week 3 in the Severity of Presence of Petechiae
Description: Percentage of subjects with change from Baseline to Week 3 in the severity of presence of petechiae was reported. Sign scores at each visit: 0= Absent, 1= Mild, 2= Moderate, 3= Severe. A decrease in score compared to baseline represented a positive outcome.
Time Frame: Baseline to Week 3
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Estriol 0.005% | Estriol 0.002% | Estriol 0.0008% | Placebo
Number analyzed (Participants) | 68 | 67 | 68 | 68
Participants
  Change from Baseline: -3 | 2 | 0 | 0 | 0
  Change from Baseline: -2 | 8 | 6 | 6 | 3
  Change from Baseline: -1 | 23 | 18 | 22 | 7
  Change from Baseline: 0 | 31 | 41 | 38 | 54
  Change from Baseline: 1 | 3 | 2 | 1 | 3
  Change from Baseline: 2 | 1 | 0 | 1 | 1
  Change from Baseline: 3 | 0 | 0 | 0 | 0
Statistical Analysis 1: Comparison: Estriol 0.005% vs Placebo; Test type: Superiority; p < 0.001, Wilcoxon rank-sum test — [p-value comment as in outcome 1, analysis 1]; Median Difference (Final Values) = 0, 95% CI 2-sided [-1 to 0] — Hodges-Lehmann estimate of location shift and corresponding asymptotic Confidence Interval
Statistical Analysis 2: Comparison: Estriol 0.002% vs Placebo; Test type: Superiority; p = 0.054, Wilcoxon rank-sum test — [p-value comment as in outcome 1, analysis 1]; Median Difference (Final Values) = 0, 95% CI 2-sided [0 to 0] — Hodges-Lehmann estimate of location shift and corresponding asymptotic Confidence Interval
Statistical Analysis 3: Comparison: Estriol 0.0008% vs Placebo; Test type: Superiority; p < 0.001, Wilcoxon rank-sum test — [p-value comment as in outcome 1, analysis 1]; Median Difference (Final Values) = 0, 95% CI 2-sided [0 to 0] — Hodges-Lehmann estimate of location shift and corresponding asymptotic Confidence Interval

27. Secondary Outcome: Change From Baseline to Week 3 in the Severity of Dry Mucosa
Description: Percentage of subjects with change from Baseline to Week 3 in severity of dry mucosa was reported. Sign scores at each visit: 0= Absent, 1= Mild, 2= Moderate, 3= Severe. A decrease in score compared to baseline represented a positive outcome.
Time Frame: Baseline to Week 3
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Estriol 0.005% | Estriol 0.002% | Estriol 0.0008% | Placebo
Number analyzed (Participants) | 68 | 67 | 68 | 68
Participants
  Change from Baseline: -3 | 4 | 8 | 6 | 3
  Change from Baseline: -2 | 29 | 20 | 26 | 17
  Change from Baseline: -1 | 22 | 30 | 21 | 20
  Change from Baseline: 0 | 12 | 9 | 15 | 26
  Change from Baseline: 1 | 1 | 0 | 0 | 2
  Change from Baseline: 2 | 0 | 0 | 0 | 0
  Change from Baseline: 3 | 0 | 0 | 0 | 0
Statistical Analysis 1: Comparison: Estriol 0.005% vs Placebo; Test type: Superiority; p = 0.008, Wilcoxon rank-sum test — [p-value comment as in outcome 1, analysis 1]; Median Difference (Final Values) = 0, 95% CI 2-sided [-1 to 0] — Hodges-Lehmann estimate of location shift and corresponding asymptotic Confidence Interval
Statistical Analysis 2: Comparison: Estriol 0.002% vs Placebo; Test type: Superiority; p = 0.01, Wilcoxon rank-sum test — [p-value comment as in outcome 1, analysis 1]; Median Difference (Final Values) = -1, 95% CI 2-sided [-1 to 0] — Hodges-Lehmann estimate of location shift and corresponding asymptotic Confidence Interval
Statistical Analysis 3: Comparison: Estriol 0.0008% vs Placebo; Test type: Superiority; p = 0.001, Wilcoxon rank-sum test — [p-value comment as in outcome 1, analysis 1]; Median Difference (Final Values) = 0, 95% CI 2-sided [-1 to 0] — Hodges-Lehmann estimate of location shift and corresponding asymptotic Confidence Interval

28. Secondary Outcome: Change From Baseline to Week 3 in Vaginal pH
Description: Change from Baseline to Week 3 in vaginal pH was reported. A decrease in pH compared to Baseline represents a positive outcome.
Time Frame: Baseline to Week 3
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: pH
Arm/Group | Estriol 0.005% | Estriol 0.002% | Estriol 0.0008% | Placebo
Number analyzed (Participants) | 68 | 67 | 68 | 68
pH | -1.03 (0.095) | -0.97 (0.096) | -0.88 (0.095) | -0.22 (0.096)
Statistical Analysis 1: Comparison: Estriol 0.005% vs Placebo; Test type: Superiority; p < 0.001, ANCOVA; LS Mean Difference = -0.81, 95% CI 2-sided [-1.071 to -0.548]
Statistical Analysis 2: Comparison: Estriol 0.002% vs Placebo; Test type: Superiority; p < 0.001, ANCOVA; LS Mean Difference = -0.75, 95% CI 2-sided [-1.013 to -0.484]
Statistical Analysis 3: Comparison: Estriol 0.0008% vs Placebo; Test type: Superiority; p < 0.001, ANCOVA; LS Mean Difference = -0.66, 95% CI 2-sided [-0.916 to -0.397]

29. Secondary Outcome: Change From Baseline to Week 3 in the Proportion of Superficial Cells of the Vaginal Epithelium
Description: Change from baseline to week 3 in the proportion of superficial cells of the vaginal epithelium was reported.
Time Frame: Baseline to Week 3
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: ratio
Arm/Group | Estriol 0.005% | Estriol 0.002% | Estriol 0.0008% | Placebo
Number analyzed (Participants) | 65 | 61 | 68 | 61
ratio | 0.48 (0.035) | 0.43 (0.036) | 0.38 (0.035) | 0.04 (0.037)
Statistical Analysis 1: Comparison: Estriol 0.005% vs Placebo; Test type: Superiority; p < 0.001, ANCOVA; LS Mean Difference = 0.44, 95% CI 2-sided [0.337 to 0.535]
Statistical Analysis 2: Comparison: Estriol 0.002% vs Placebo; Test type: Superiority; p < 0.001, ANCOVA; LS Mean Difference = 0.39, 95% CI 2-sided [0.291 to 0.494]
Statistical Analysis 3: Comparison: Estriol 0.0008% vs Placebo; Test type: Superiority; p < 0.001, ANCOVA; LS Mean Difference = 0.34, 95% CI 2-sided [0.245 to 0.439]

30. Secondary Outcome: Change From Baseline to Week 3 in the Proportion of Parabasal Cells of the Vaginal Epithelium
Description: Change from Baseline to Week 3 in the proportion of parabasal cells of the vaginal epithelium was reported. A decrease in proportion of parabasal cells compared to baseline represents a positive outcome.
Time Frame: Baseline to Week 3
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: ratio
Arm/Group | Estriol 0.005% | Estriol 0.002% | Estriol 0.0008% | Placebo
Number analyzed (Participants) | 65 | 61 | 68 | 61
ratio | -0.55 (0.037) | -0.57 (0.037) | -0.48 (0.036) | -0.08 (0.038)
Statistical Analysis 1: Comparison: Estriol 0.005% vs Placebo; Test type: Superiority; p < 0.001, ANCOVA; LS Mean Difference = -0.47, 95% CI 2-sided [-0.575 to -0.371]
Statistical Analysis 2: Comparison: Estriol 0.002% vs Placebo; Test type: Superiority; p < 0.001, ANCOVA; LS Mean Difference = -0.49, 95% CI 2-sided [-0.592 to -0.383]
Statistical Analysis 3: Comparison: Estriol 0.0008% vs Placebo; Test type: Superiority; p < 0.001, ANCOVA; LS Mean Difference = -0.4, 95% CI 2-sided [-0.5 to -0.3]

ADVERSE EVENTS:
Time Frame: Adverse events were assessed from the time the subject signed the ICF until exit from the study, aproximately 20 weeks
Description: The safety population included all randomized subjects who received at least 1 dose of study treatment. Data for treatment-emergent adverse events is presented here. Subjects were questioned and observed for evidence of AEs. For any preexisting condition or abnormal laboratory finding that changed in severity after dosing, the change was to be recorded as an AE. New abnormal laboratory findings that were considered clinically significant by the Investigator were considered AEs.
Arm/Group | Estriol 0.005% | Estriol 0.002% | Estriol 0.0008% | Placebo
All-Cause Mortality (participants affected / at risk) | 0/70 | 0/69 | 0/72 | 0/71
Serious Adverse Events (participants affected / at risk) | 0/70 | 0/69 | 0/72 | 3/71
Other Adverse Events (participants affected / at risk) | 14/70 | 11/69 | 15/72 | 20/71
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Estriol 0.005% (N=70) | Estriol 0.002% (N=69) | Estriol 0.0008% (N=72) | Placebo (N=71)
Non-Hodgkin´s lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — The event started 7 months after the subject completed the study
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Estriol 0.005% (N=70) | Estriol 0.002% (N=69) | Estriol 0.0008% (N=72) | Placebo (N=71)
Flushing (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Breast inflammation (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ovarian cyst (Reproductive system and breast disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Vulvovaginal burning sensation (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vulvovaginal pruritus (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Accidental overdose (Injury, poisoning and procedural complications) | 4 (5) | 3 (4) | 4 (4) | 3 (4)
Animal bite (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neck injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Radius fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood glucose increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Flatulence (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperchlorhydria (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Loose tooth (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Leukocyturia (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Arthritis reactive (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperuricaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bacterial vaginosis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cystitis (Infections and infestations) | 0 (0) | 1 (1) | 2 (3) | 3 (3)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 0 (0) | 1 (1) | 1 (2) | 1 (1)
Nasopharyngitis (Infections and infestations) | 1 (1) | 2 (2) | 3 (3) | 3 (3)
Pharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tooth abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 3 (3)
Viral infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Vulval abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Statistical Analysis Plan (2017-06-22): https://cdn.clinicaltrials.gov/large-docs/10/NCT02967510/SAP_000.pdf
  • Study Protocol (2017-06-07): https://cdn.clinicaltrials.gov/large-docs/10/NCT02967510/Prot_001.pdf